CLINICAL TRIAL: NCT06650306
Title: The Impact of Soft Contact Lenses on the Corneal Neuromediators and Optical Quality in High Myopia Prior to SMILE
Status: Recruiting | Type: Observational
Sponsor: yuhao shao (Other)
Responsible Party: Sponsor-Investigator, yuhao shao, MD, Tongji University
Organization: Tongji University (Other)
Other Study IDs: SHSY-IEC-5.0/23K74/P01
Record Dates: First submitted 2024-10-16; First posted 2024-10-21 (Actual); Last update posted 2024-10-21 (Actual); Status verified 2024-10

CONDITIONS: Contact Lens Complication
Keywords: Corneal Neuromediator; Soft contact lenses; Corneal optical density; Corneal aberration

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Biospecimen Retention: Samples With DNA — All samples were collected from participants with high myopia who underwent SMILE surgery. The VisuMax femtosecond laser system (Carl Zeiss Meditec, Jena, Germany) was utilized with the following settings: a repetition rate of 500 kHz, pulse energy of 150 nJ, intended cap thickness of 110-120 μm, and optical zone of 6.0-6.8 mm. A circumferential incision width of 2 mm was made for lenticule dissection and extraction. The surgical procedures were performed by a single experienced surgeon (Dr. Zou). Following the SMILE surgeries, corneal stromal lenticules were transferred to Eppendorf tubes and stored at -80°C. for subsequent analysis.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (3):
- SCLs >10 years: high myopia patients who wear SCL more than 10 years before Small Incision Lenticule Extraction
  Interventions: Other: This study does not involve any interventions
- SCLs ≤10 years: high myopia patients who wear SCL for 10 years or less before Small Incision Lenticule Extraction
  Interventions: Other: This study does not involve any interventions
- NW: high myopia patients who have not worn SCLs before Small Incision Lenticule Extraction
  Interventions: Other: This study does not involve any interventions

INTERVENTIONS:
Other: This study does not involve any interventions — This study does not involve any interventions

SUMMARY:
To investigate the influence of Neuromediators expression in corneal stromal lenticules and corneal injury repair after small incision extraction

DETAILED DESCRIPTION:
This study included 160 eyes from high myopia patients who underwent Small Incision Lenticule Extraction. Patients were devided into three groups based on duration of wearing SCLs: > 10 years group, ≤ 10 years group, and NW group (not SCLs). Corneal higher-order aberrations and densitometry were evaluated using a Pentacam system. Neuromediator levels in corneal stromal lenticules were analyzed using ELISA and immunofluorescence

ELIGIBILITY:
Inclusion Criteria:

* age ≥ 18 years with stable refraction for at least two years;
* spherical equivalent (SE) < -6.00 D;
* corrected distance visual acuity of 20/20 or better;
* no history of using rigid gas permeable lenses or orthokeratology (OK) lenses prior to examination

Exclusion Criteria:

- a history of moderate to severe dry eye as well as any ocular or systemic disease that would contraindicate laser refractive surgery.

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: patients with high myopia who underwent SMILE surgery at Shanghai Tenth People's Hospital in Shanghai, China, between October 2020 and October 2023.
Sampling Method: Non-Probability Sample
Enrollment: 80 (Estimated)
Dates: Start 2024-10-18 (Actual); Primary Completion 2026-06-30 (Estimated); Study Completion 2026-06-30 (Estimated)

PRIMARY OUTCOMES:
Corneal stromal lenticule Neuromediators | baseline
  Corneal neuromediators, including NGF(pg/mL), CGRP(pg/mL), SP(pg/mL), IGFBP-1(ng/mL), and MANF(pg/mL), which play pivotal roles in maintaining normal physiological functions of the cornea.

SECONDARY OUTCOMES:
Corneal Aberration | baseline
  Preoperative corneal aberration measurements were performed using a Scheimpflug tomography system (Pentacam; Oculus GmbH, Wetzlar, Germany). Images of the highest quality (designated as OK) were selected for analysis. The coefficients for a standardized diameter of 8 ?mm were examined, followed by an assessment of the clinical significance of total higher-order aberrations (HOA, mm), spherical aberration (Z4, 0, mm), horizontal coma (Z3, 1, mm), vertical coma (Z3, -1, mm), horizontal trefoil (Z3, 3, mm), and oblique trefoil (Z3, -3, mm) in relation to visual quality.
Corneal Densitometry | baseline
  The Pentacam HR was used to collect data on corneal densitometry values, which were expressed in grayscale units (GSUs), playing a crucial role in quantifying corneal clarity by monitoring transient haze-like reactions. The cornea was divided into four annular zones (0-2 mm, 2-6 mm, 6-10 mm, and 10-12 mm), each exhibiting distinct corneal densitometry values. Based on the anatomical layers of the cornea at different depths, it consists of four layers: a superficial anterior layer of 120 μm, a posterior layer located within the innermost part of the cornea measuring 60 μm; central layers calculated by subtracting thickness of the anterior and posterior layers from the total layer thickness; and a total layer. Corneal densitometry values were measured in the 0-2 mm and 2-6 mm to correspond to the corneal optical zone diameter of SMILE.

CONTACTS AND LOCATIONS:
Locations (1):
- Shanghai Tenth People's Hospital, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: No